CLINICAL TRIAL: NCT05470140
Title: A Phase 1 Study of WU-NK-101 in Patients With Relapsed or Refractory (R/R) Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wugen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WUN101-01
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: relapsed, refractory, leukemia, NK cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia

STUDY DESIGN:
Intervention Model Description: This study will determine the safety and tolerability of WU-NK-101 and define the RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: WU-NK-101 (Experimental): A non-engineered Natural Killer (NK) cell derived from peripheral blood mononuclear cells (PBMC) that is cytokine-reprogrammed, expanded, and cryopreserved to create an allogeneic enhanced Memory-like anti-tumor NK cell therapy product.
  Each 28-day cycle of treatment consists of 3 doses of WU-NK-101 administered on Day 1, Day 8, and Day 15.
  Interventions: Biological: WU-NK-101

INTERVENTIONS:
Biological: WU-NK-101 — WU-NK-101 administered on Day 1, Day 8, and Day 15.

SUMMARY:
This study is a Phase 1, open-label, dose escalation, and cohort expansion study designed to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary anti-leukemic activity of WU-NK-101 in R/R AML.

DETAILED DESCRIPTION:
This is a first in human, multi-center Phase 1 single agent study in patients with R/R AML who have exhausted other treatment options. The study will consist of two phases, dose escalation and cohort expansion. During the Dose Escalation Phase, up to 18 patients will be treated with WU-NK-101 in up to 3 Dose Levels (DL) until maximum tolerated dose (MTD) or maximum administered dose (MAD) is determined.

Once the MTD/MAD is defined, 6 additional patients will be enrolled in the Cohort Expansion Phase to further characterize the safety, tolerability, as well as determining the recommended phase 2 dose (RP2D) of WU-NK-101. Patients in the Cohort Expansion Phase, who achieve a partial response (PR), may receive up to 2 further re-induction cycles contingent on safety in the Dose Escalation Phase; patients who achieve a complete remission with partial hematologic recovery (CRh) or complete remission with incomplete hematologic recovery (CRi) at any point during the course of treatment may receive a further consolidation cycle, for a total of up to 4 cycles per patient. During cohort expansion, dosing breaks of up to two weeks are allowed between cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of primary or secondary AML (any subtype except acute promyelocytic leukemia) according to World Health Organization (WHO) 2016 classification
2. Unlikely to benefit from standard of care therapy
3. Patients with AML post hematopoietic stem cell transplant (HSCT) [permitted in Cohort Expansion Phase only] must meet the following criteria:

   * There must be histological confirmation of AML relapse after HSCT
   * Undergone allogeneic HSCT (alloSCT) > 90 days prior to enrollment from a match related donor, matched unrelated donor, cord blood donor, or haplo- identical donor
   * Off all immunosuppressive medications for a minimum of 2 weeks
4. Adequate organ function as defined in the protocol
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2 at screening

Exclusion Criteria:

1. Circulating blast count >30,000/µL by morphology or flow cytometry (cytoreductive therapies such as leukapheresis or hydroxyurea are allowed)
2. Uncontrolled or untreated bacterial, fungal, or viral infections, including HIV, Hepatitis B or C infection, or uncontrolled infection of any etiology
3. Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiogram (ECG) suggestive of acute ischemia or active conduction system abnormalities
4. Severe renal impairment, defined as creatinine clearance <40 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events of WU-NK-101 as assessed by CTCAE v5 | 24 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of consent until End of Study (EOS) visit.
Maximum Tolerated Dose | Up to 21 days from first dose
  Maximum Tolerated or Administered Dose of WU-NK-101

SECONDARY OUTCOMES:
Overall Survival | 3 months
  Time from study drug administration (Day 1) until death on study.
Duration of Response | 24 months
  Time of response to the time of disease relapse, progression, or death due to any cause.
Overall Response Rate (ORR) | 24 months
  ORR is defined as proportion of patients that achieve complete remission (CR) + complete remission with incomplete hematologic recover (CRi).

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Thomas, MD, Study Director — Wugen, Inc.
Locations (9):
- United States (6):
  - City of Hope, Duarte, California
  - Stanford Healthcare, Palo Alto, California
  - Norton Health Care, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Providence Portland Medical Center, Portland, Oregon
- Australia (3):
  - Peter MacCallum Cancer Center, Melbourne
  - Royal Perth Hospital, Perth
  - Royal Prince Alfred Hospital, Sydney